CLINICAL TRIAL: NCT01792180
Title: The Senior Step Study: How Elderly Help Themselves Maximally Forward
Brief Title: The Senior Step Study How Elderly Help Themselves Maximally Forward
Acronym: SSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Marcel Olde Rikkert, Prof dr, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Nr. 60-61900-98-449
Record Dates: First submitted 2013-02-11; First posted 2013-02-15 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Self-management for Mobility Improvement in the Elderly
Keywords: Gait speed; Mobility; Falls; Fall risk; Self-management; Mental wellbeing; Elderly

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): No intervention besides weekly telephone calls from the computerized falls telephone system
- Intervention group (Experimental): Weekly use of the mobility feedback device, use of instruction book with every day exercises, use of activity diary in intervention group.
  Interventions: Behavioral: Mobility feedback device with use of instruction book

INTERVENTIONS:
Behavioral: Mobility feedback device with use of instruction book — Weekly use of the mobility feedback device to measure gait speed. Two infrared sensors will be placed in the line of walking, a photo frame containing a display, symbols and lights will tell the participant when and how to perform the test. Gait speed is shown on the display and will serve as feedback to the participant. Participant can use their gait speed to decide which exercises from the instruction book he performs. Participants will be asked to keep an activity diary.
  Arms: Intervention group

SUMMARY:
The Senior Step Study investigates whether feedback given by a mobility feedback device in combination with an instruction book containing every day exercises, motivates elderly to exercise more. By exercising more participants take charge of their own mobility and fall risk. Senior Step Study studies whether this 'exercising more' positively affects their mobility, fall risk, mental wellbeing, self-management, and quality of life.

DETAILED DESCRIPTION:
Falling is an important problem among community-dwelling elderly. The number of falls and concomitant health costs will rise within an aging population. Fall related injuries and fear of falling decrease mobility and have a negative impact on social functioning, mood, wellbeing and autonomy. Research from a medical perspective has concentrated on case finding and fall prevention. Currently, insufficient possibilities are available for elderly and caregiver to asses and improve their own mobility and fall risk. The Senior Step Study aims to provide a tool for elderly to improve their self-management abilities in monitoring and improving mobility and fall risk.

The researchers expect that elderly in the intervention group will be more aware of their own mobility and fall risk, and will therefore experience more autonomy, better mental wellbeing, and better quality of life. We expect this to reflect in less demands made on healthcare by the elderly.

150 elderly living at home, in a home for the elderly, and elderly who regularly attend activities in a community home, are asked to participate in the study. During the six months of the study, subjects will receive weekly telephone calls from the computerized falls telephone. The intervention group will measure their normal gait speed measured over 4 meters, using the mobility feedback device once a week, and use the feedback given by this mobility feedback device to perform exercises from the instruction book. Activity diaries allow them to register the type and duration of the exercises.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of 70 years and over
* Subjects who experienced at least 1 fall in the previous 12 months
* Subjects who can walk independently or with a walking aid
* Informed consent on the basis of Dutch legislation (WMO)
* During the study subjects cannot participate in a falls prevention course

Exclusion Criteria:

* Subjects not able to speak Dutch
* Subjects not able to understand and remember simple Dutch instructions
* Subjects not capable of using the falls telephone, and do not have an informal caregiver who can answer the falls telephone for them

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Mental wellbeing | Baseline to 3 months
  Medical Outcomes Study (MOS-20)

SECONDARY OUTCOMES:
Number of falls | Baseline to 6 months
  Computerized falls telephone system
Self-management | Baseline to 3 months, baseline to 6 months
  Self-Management Ability Scale (SMAS-30)
Physical activity | Baseline to 3 months, baseline to 6 months
  LASA Physical Activity Questionnaire (LAPAQ)
Fear of falling | Baseline to 3 months, baseline to 6 months
  Falls Efficacy Scale (FES-I)
Balance and mobility | Baseline to 3 months, baseline to 6 months
  Short Physical Perfomance Battery, Timed Up and Go
Mental Wellbeing | Baseline to 6 months
  Medical Outcomes Study (MOS-20)

OTHER OUTCOMES:
Compliance and motivation using the intervention | Baseline to 6 months
  Qualitative research using semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Marcel GM Olde Rikkert, Prof PhD MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
raw data can be shared